CLINICAL TRIAL: NCT04175093
Title: A Study on Some Biomarkers in Bronchial Asthma in Children
Brief Title: Some Biomarkers in Bronchial Asthma in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Sara Safwat Abd-Elaleem Hafez, Principal investigator, Assiut University
Other Study IDs: BRASTHMA
Record Dates: First submitted 2019-11-20; First posted 2019-11-22 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild persistent asthma: • Group I, patients with mild persistent asthma.
  Interventions: Diagnostic Test: asymmetric dimethylarginine
- Moderate persistent asthma: • Group II, patients with moderate persistent asthma.
  Interventions: Diagnostic Test: asymmetric dimethylarginine
- Severe persistent asthma: • Group III ,patients with severe persistent asthma.
  Interventions: Diagnostic Test: asymmetric dimethylarginine

INTERVENTIONS:
Diagnostic Test: asymmetric dimethylarginine — measurement by ELISA of asymmetric dimethylarginine

SUMMARY:
Asthma, a disease characterized by chronic airway inflammation and hyper -responsiveness, is a common disease that affects all age groups. Asthma may be manifested as irreversible airflow obstruction in some patients. Although the pathogenesis of asthma is not well understood, increased oxidative stress due to an imbalance of oxidants and antioxidants has been found to be associated with asthma. In asthma, inflammation-related oxidative stress is driven by exposure to a variety of triggers, including allergens and viruses, which activate components of both the innate and acquired immune responses. Protection by escaping from triggering factors or standardization of asthma medication is difficult and usually is not enough for effective treatment. On the other hand, correction of antioxidative systems may be more efficacious in the control of asthmatic inflammation and asthma symptoms.

Little is known about the role of asymmetric dimethylarginine in the pathogenesis of asthmatic airway inflammation. The lung is a major source of asymmetric dimethylarginine that can promote oxidative stress by a reduction in nitric oxide synthesis which would result in higher levels of peroxynitrite, that causes oxidative cell damage, and exacerbate airway inflammation. asymmetric dimethylarginine can modify lung function, increase airway hyper-reactivity even in non-inflamed airways, and promote lung collagen production and deposition. Increased asymmetric dimethylarginine in serum has been found to be associated with the severity of symptoms of asthma in obese adults.

Malondialdehyde is an oxidant marker of pulmonary oxidative stress, and lipid peroxidation. Paraoxonase, an antioxidant enzyme may play a protective role in asthma. It hydrolyzes lipid peroxides and prevents low-density lipoprotein oxidation.

ELIGIBILITY:
• All known asthmatic patients aged six years or more who will be regularly attending Assuit University Children's Hospital Outpatient clinic.

Exclusion criteria include

* Obese children,
* The presence of chronic heart, liver and kidney diseases, concomitant chronic inflammatory disease and autoimmune disorders, and Diabetes mellitus.
* Patients taking antioxidant drugs, vitamins, diuretics, hormone replacement therapy will be also excluded.
* Children aged less than six years. 5-children who have symptoms of lower or upper respiratory tract infection or asthma exacerbation within the previous four weeks.

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All the children included in the study will be exposed to full clinical examination and history for assessment of severity of asthma in patient groups according to the guidelines for diagnosis and managemt of asthma 2007.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2019-11-29 (Estimated); Primary Completion 2020-11-21 (Estimated); Study Completion 2021-11-21 (Estimated)

PRIMARY OUTCOMES:
The percentage of asymmetric dimethylarginine in the study groups | 24 hours
  measurement from serum samples by competitive ELISA with a standard range from 0.1 to 5.0 μmol/L.

IPD SHARING:
Plan to Share IPD: No